CLINICAL TRIAL: NCT02430909
Title: A Double-blind, Randomized, Placebo-controlled Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of Multiple Doses of UCB4940 Administered as Add-on to Certolizumab Pegol Therapy in Subjects With Moderate-to-Severe Rheumatoid Arthritis
Brief Title: Multiple Dose Study of UCB4940 as add-on to Certolizumab Pegol in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Celltech (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA0123; 2014-003307-30 (EudraCT Number)
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — bimekizumab; Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CZP / CZP + PBO / CZP (Placebo Comparator): Certolizumab Pegol (400 mg at Weeks 0, 2, and 4 followed by 200 mg every two weeks) until Week 30
  +Placebo from Week 8 to Week 18
  Interventions: Biological: Certolizumab Pegol; Other: Placebo
- CZP / CZP + UCB4940 / CZP (Experimental): Certolizumab Pegol (400 mg at Weeks 0, 2, and 4 followed by 200 mg every two weeks) until Week 30
  + UCB4940 from Week 8 until Week 18
  Interventions: Biological: Bimekizumab; Biological: Certolizumab Pegol
- CZP / CZP/ CZP (Other): Certolizumab Pegol (400 mg at Weeks 0, 2, and 4 followed by 200 mg every two Weeks) until Week 30
  Interventions: Biological: Certolizumab Pegol

INTERVENTIONS:
Biological: Bimekizumab — * Pharmaceutical form: Solution for infusion
  * Concentration: Vials at 80 mg/ml will be diluted with 0.9% sodium chloride to a final concentration to achieve the correct dose
  * Route of administration: iv infustion
  Arms: CZP / CZP + UCB4940 / CZP
Biological: Certolizumab Pegol — * Pharmaceutical form: Prefilled syringes
  * Concentration: 200 mg/ml
  * Route of administration: Subcutaneous injection
Other: Placebo — * Pharmaceutical form: Solution for infusion
  * Concentration: 0.9% saline
  * Route of administration: Intravenous infusion
  Arms: CZP / CZP + PBO / CZP

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and body distribution of Bimekizumab (UCB4940) when added to Certolizumab Pegol treatment in patients with Rheumatoid Arthritis. Neither the patient nor the doctor will know the treatment group.

ELIGIBILITY:
Inclusion Criteria

To be eligible to participate in this study, all of the following criteria must be met:

* Subject is informed and given approved written Informed Consent Form (ICF).
* Subject is considered reliable and capable of adhering to the protocol.
* Subject must have a diagnosis of adult-onset moderate-to-severe RA of at least 6 months' duration as defined by ACR/EULAR 2010 classification criteria.
* Subject must have:

  * ≥6 tender joints (out of 68)
  * ≥6 swollen joints (out of 66)
  * CRP≥10.0mg/L .
* Subject must have had inadequate response to at least 1 synthetic DMARD.
* Subject is at least 18 years and less than 70 years of age at Visit 1 (Screening).
* Female subjects must either be:

  * postmenopausal
  * permanently sterilized or,
  * if of childbearing potential, must be willing to use at least 2 effective methods of contraception,
* Male subjects with partners of childbearing potential must be willing to use a condom when sexually active, during the study and for 5 months after last administration of study drug.

Exclusion Criteria

Subjects are not permitted to enroll in the study if any of the following criteria is met:

* Subject has previously participated in this study or has previously been assigned to treatment in a study of the investigational medicinal product (IMP) under investigation in this study (UCB4940 and/or CZP).
* Subject has a history or active systemic/respiratory infection due to fungal, parasitic, or mycotic pathogens.
* Subjects with known tuberculosis (TB) infection, at high risk of acquiring TB infection, or latent TB infection are excluded.
* Subject is at high risk of infection.
* Subject has an active infection or has had a serious infection within 12 weeks prior to the first dose of study drug at Week 0.
* Subject has renal or liver impairment.
* Subject has a current or past history of gastrointestinal ulceration.
* Subject has active neoplastic disease or history of neoplastic disease.
* Subject has a concomitant diagnosis of any other inflammatory condition.
* Subject has a secondary, non-inflammatory condition or a known diagnosis of fibromyalgia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Screening (D-28) until final study visit (Week 44)
  All adverse events (AEs) are recorded during the entire study period.
Change from Baseline 2 in DAS28(CRP) | Week 20
  DAS28 (Disease Activity Score 28) is a measure of disease activity in Rheumatoid Arthritis (RA) and is a composite score derived from the number of swollen and tender joints (out of 28), the CRP value and the patient global assessment of disease activity.

SECONDARY OUTCOMES:
Percent improvement in ACR (American College of Rheumatology) criteria (ACRn) based on Baseline 2 | Week 20
  ACRn is the percentage improvement from Baseline 2 in the number of tender joints, in the number of swollen joints, and in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
ACR20 response based on Baseline 2 | Week 20
  The assessments are based on a 20% or greater improvement from Baseline 2 in the number of tender joints, in the number of swollen joints, and a 20% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
ACR50 response based on Baseline 2 | Week 20
  The assessments are based on a 20% or greater improvement from Baseline 2 in the number of tender joints, in the number of swollen joints, and a 50% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
ACR70 response based on Baseline 2 | Week 20
  The assessments are based on a 20% or greater improvement from Baseline 2 in the number of tender joints, in the number of swollen joints, and a 70% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
DAS28(CRP) remission | Week 20
  DAS28(CRP) remission is defined as DAS28(CRP) < 2.6. DAS28 is a measure of disease activity in RA and is a composite score derived from the number of swollen and tender joints (out of 28) , the C-reactive protein value and the patient global assessment of disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (21):
- Ra0123 101, Prague, Czechia
- Hungary (4):
  - Ra0123 203, Balatonfüred
  - Ra0123 201, Budapest
  - Ra0123 202, Budapest
  - Ra0123 204, Budapest
- Ra0123 801, Chisinau, Moldova
- Poland (5):
  - Ra0123 303, Bialystok
  - Ra0123 306, Lublin
  - Ra0123 304, Poznan
  - Ra0123 305, Poznan
  - Ra0123 301, Warsaw
- Russia (8):
  - Ra0123 403, Moscow
  - Ra0123 404, Moscow
  - Ra0123 405, Moscow
  - Ra0123 406, Moscow
  - Ra0123 408, Moscow
  - Ra0123 407, Saint Petersburg
  - Ra0123 402, Yaroslavl
  - Ra0123 410, Yaroslavl
- Ra0123 501, Bratislava, Slovakia
- Ra0123 601, Glasgow, United Kingdom

REFERENCES:
- [Derived] Glatt S, Taylor PC, McInnes IB, Schett G, Landewe R, Baeten D, Ionescu L, Strimenopoulou F, Watling MIL, Shaw S. Efficacy and safety of bimekizumab as add-on therapy for rheumatoid arthritis in patients with inadequate response to certolizumab pegol: a proof-of-concept study. Ann Rheum Dis. 2019 Aug;78(8):1033-1040. doi: 10.1136/annrheumdis-2018-214943. Epub 2019 Jun 8. PMID 31177099